CLINICAL TRIAL: NCT07272148
Title: The Pilot of the Turku Outpatient Clinic for Functional and Fatigue Disorders in the Welbeing Services County of Southwest Finland
Brief Title: The Pilot of the Turku Outpatient Clinic for Functional and Fatigue Disorders
Acronym: TOCliFFD
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T1398-2023-2
Record Dates: First submitted 2025-11-17; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Persistent Physical Symptoms (PPS); Functional Disorder; Fatigue Syndrome, Chronic
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering persistent symptoms: The clinic's staff included a pilot project coordinator, a physician, an occupational therapist, a physiotherapist, a psychologist, a rehabilitation counselor, and a ward secretary. At the physician's initial visit, stress system sensitization, burden factors, and need for symptomatic medication were assessed. In a joint rehabilitation team meeting, the patient met a psychologist, occupational therapist, physiotherapist, and rehabilitation counselor, who conducted a multidisciplinary evaluation and created an individualized rehabilitation plan. Patients then attended a course for persistent bodily symptoms, with some joining a psychophysical breathing group. Individual rehabilitation or counseling was provided according to each patient's needs.
  Interventions: Behavioral: Biopsychosocial, multidisciplinary, and individually tailored rehabilitation for patients with persisten symptoms

INTERVENTIONS:
Behavioral: Biopsychosocial, multidisciplinary, and individually tailored rehabilitation for patients with persisten symptoms — The clinic's staff included a pilot project coordinator, a physician, an occupational therapist, a physiotherapist, a psychologist, a rehabilitation counselor, and a ward secretary. At the physician's initial visit, stress system sensitization, burden factors, and need for symptomatic medication were assessed. In a joint rehabilitation team meeting, the patient met a psychologist, occupational therapist, physiotherapist, and rehabilitation counselor, who conducted a multidisciplinary evaluation and created an individualized rehabilitation plan. Patients then attended a course for persistent bodily symptoms, with some joining a psychophysical breathing group. Individual rehabilitation or counseling was provided according to each patient's needs.

SUMMARY:
This study examined 125 working-age patients from the Turku Outpatient Clinic for Functional and Fatigue Disorders. "Patients participate in the clinic's biopsychosocial, multidisciplinary, and individually tailored rehabilitation. The aim of the rehabilitation is to improve patients' functional capacity and provide them with tools to manage and cope with their symptoms. In addition, the goal is to break the cycle of unnecessary examinations that cause harm to the patient. Socioeconomic data, as well as information related to functional capacity, symptoms, and quality of life, are collected from patients at the start of rehabilitation and again at six and twelve months after the beginning of rehabilitation. In addition, data on patients' use of social and health care services are requested from registers for the year preceding the start of rehabilitation and for the year following rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering persistent symptoms
* referred to the clinic between August 1, 2023 to April 30, 2025

Exclusion Criteria:

* ineligible for the study because of the need for extensive additional examinations in a specialized field, acute substance abuse problems, and/or lack of motivation.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of working-age patients with persistent symptoms in the wellbeing services county of Southwest Finland. Referrals to the clinic were made from primary health care, occupational health care, private health services, and specialized health care.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quality of life of the patients | At baseline and at 6 and 12 months follow-ups
  WHOQOL-BREF

SECONDARY OUTCOMES:
Functional limitations of the patients | At baseline and at 6 and 12 months follow-up
  WHODAS 2.0

OTHER OUTCOMES:
Use of social and health services | At baseline and at 6 and 12 month follow-ups
  Number of visits and service fee per visits

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Health and Social Services Centre, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Only upon reasonable request.